CLINICAL TRIAL: NCT02324556
Title: A LAparoscopic and TransAnal Total Mesorectal Excision (TME for Rectal Cancer Trial
Brief Title: A LAparoscopic and TransAnal Total Mesorectal Excision (TME) for Rectal Cancer Trial
Acronym: LATA
Status: Terminated | Type: Observational
Why Stopped: Patients are currently being operated in the robot instead due to logistics
Sponsor: Sahlgrenska University Hospital (Other)
Responsible Party: Principal Investigator, Eva Angenete, Senior Consultant Surgeon, Associate professor, Sahlgrenska University Hospital
Other Study IDs: LATA
Record Dates: First submitted 2014-11-27; First posted 2014-12-24 (Estimated); Last update posted 2020-04-28 (Actual); Status verified 2020-04

CONDITIONS: Colorectal Neoplasm
Keywords: Rectal Cancer; Surgery; Laparoscopy
MeSH Terms: conditions — Colorectal Neoplasms; Rectal Neoplasms

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Laparoscopic total mesorectal excision: Patients operated with laparoscopic total mesorectal surgery for rectal cancer
- transanal total mesorectal excision: Patients operated with a combined transanal and laparosocopic total mesorectal surgery for rectal cancer

SUMMARY:
All patients planned for an anterior resection due to rectal cancer with a total mesorectal excision are included. This is a feasibility study, thus no randomization will be performed.

Primary endpoint is clinical and pathologic examination of the specimen. Secondary end-points include clinical variables such as conversion rate, re-admission and/or re-operation due to any complication and health economy analyses.

DETAILED DESCRIPTION:
The design is comparative and prospective, we will compare specimens from patients operated at our institution during the last year with standard open or laparoscopic approach with patients operated with the new technique. Patients in the control arm will be patients operated prior to the commencement of the new technique or patients not eligible or possible to include in the study.

It is possible to obtain a macroscopically and microscopically adequate specimen after a combined approach with laparoscopic and transanal TME compared to open or laparoscopic conventional TME.

ELIGIBILITY:
Inclusion Criteria:

* presenting with a rectal cancer possible to operate with a total mesorectal excision and an anastomosis according to the local multidisciplinary conference
* possible to operate with laparoscopic technique
* possible to operate in regard to concomitant disease
* giving informed consent to participate

Exclusion Criteria:

-Participation in other trials in conflict with the protocol and end-points the LATA-trial

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Rectal cancer possible to operate with an anterior resection.
Sampling Method: Non-Probability Sample
Enrollment: 6 (Actual)
Dates: Start 2015-01; Primary Completion 2015-06 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
Number of specimens with grade I specimen according to Quirke | 4 weeks postoperatively
  Comparison with control group

SECONDARY OUTCOMES:
Conversion rate | day of surgery
Re-admission | 30 days
Postoperative complications scored according to Clavien-Dindo within the first 12 months | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Eva Angenete, M.D., Ph.D., Principal Investigator — Sahlgrenska Universitetssjukhuset/Östra
Locations (2):
- Sweden (2):
  - Dept. of Surgery, Sahlgrenska University Hospital/Ostra, Gothenburg
  - NU-sjukvården, Trollhättan